CLINICAL TRIAL: NCT01098890
Title: Intraventricular Tissue Plasminogen Activator in the Management of Aneurysmal Subarachnoid Hemorrhage: a Randomized Controlled Pilot Study
Brief Title: Intraventricular Tissue Plasminogen Activator (tPA) in the Management of Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Dr. Andreas Kramer, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22461
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-04

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Intraventricular Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be administered every 12 hours for a total five doses. Patients will be followed for a total of 6 months.
  Interventions: Drug: Placebo
- tPA (tissue plaminogen activator) (Active Comparator): Intraventricular TPA will be administered every 12 hours for a total five doses. Patients will be followed for a total of 6 months.
  Interventions: Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Tissue Plasminogen Activator — 2mg tPA will be given every twelve hours for a maximum of 5 doses
  Other Names: Cathflo
  Arms: tPA (tissue plaminogen activator)
Drug: Placebo — Placebo will be administered every 12 hours for a maximum of 5 doses.
  Arms: Placebo

SUMMARY:
The proposed study is to evaluate the acceleration the clearance of intraventricular blood (IVH) and subarachnoid hemorrhage (SAH) following ruptured intracranial aneurysms, thereby ameliorating complications, such as cerebral vasospasm, hydrocephalus and intracranial hypertension.

The primary objectives are:

1. Estimate the rate and variance of hematoma clearance following aneurysmal SAH, thereby facilitating sample size determination for a subsequent larger study;
2. Assess the feasibility of a randomized controlled trial of intraventricular tissue plasminogen activator (TPA) among patients with SAH (enrollment rate, ability to blind investigators, protocol compliance);
3. Confirm the safety of intraventricular TPA.

DETAILED DESCRIPTION:
Outcome Measures:

Safety will be assessed through adverse events, hemorrhagic complications and the development of ventriculostomy-related infections.

The volume and clearance of intracranial blood will be determined (in ml) using computerized software, as well as validated semi-quantitative ordinal scales (SAH Sum Score, Modified Graeb Score). The amount of IVH and SAH will be assessed at baseline (day 0), 72 hours after treatment onset, and on post-SAH day 8.

Additional secondary outcomes will include:

1. The occurrence of vasospasm, as determined using transcranial Doppler ultrasonography
2. The occurrence of radiographic vasospasm, using CT angiography.
3. The occurrence of "clinical" (symptomatic) vasospasm
4. The rate of catheter-related central nervous system infections
5. Levels of cytokines, endothelin and matrix metalloproteases in cerebrospinal fluid (CSF) and plasma
6. Levels of fibrin-derived products (FDP), TPA and plasminogen-activator inhibitor in CSF
7. Levels of S100β and neuron-specific enolase (NSE) in CSF and serum
8. Intracranial pressure
9. Volume of CSF drainage
10. Extended Glasgow Outcome Scale, modified Rankin scale, EuroQOL at 6 months post-SAH
11. Duration that ventriculostomy is required; need for permanent shunt
12. Fever burden

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old) with a proven ruptured cerebral aneurysm
* Aneurysm has been / will be treated with coil embolization
* EVD has been / will be placed as part of routine care
* Modified Fisher score is 4 (cisternal blood > 1 mm thick with concomitant IVH)
* CT scan after EVD placement shows "stability" with no increase in the amount of intracranial blood (Note: there is sometimes layering of blood, especially in the occipital horns of the lateral ventricles, that develops during the first 24-48 hours after a ruptured aneurysm due to circulation of blood in the CSF - this does not necessarily constitute an exclusion criterion).
* Study drug can be administered within 72 hours of the time of SAH.

Exclusion Criteria:

* Concern expressed by endovascular neurosurgeon / interventional radiologist that aneurysm has only been incompletely treated / isolated by coil embolization.
* Patient requires craniotomy and clipping of the culprit aneurysm.
* CT scan performed post-EVD insertion OR post-coiling shows increase in amount of intracranial blood.
* Uncorrected coagulation disturbance (INR > 1.5, PTT > 45); correction is permitted (if coagulation disturbance develops during the study, subsequent doses of TPA should simply be withheld until coagulation can be corrected).
* Uncorrected thrombocytopenia (platelets < 50,000); correction with platelet transfusions is permitted.
* Involvement in another clinical trial
* Uncontrolled active internal hemorrhage
* Known allergy to study drug
* Patient is pregnant
* Any other condition the investigator believes would place the subject at risk if included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Determine rate and variance of ventricular and cisternal clot clearance (with and without TPA). | 8 Days post bleed
  In order to plan the sample size for a future "proof-of-concept" trial, we need to better define the primary endpoint (the rate of ventricular and cisternal clot clearance, as well as the degree of variance in this rate, both with and without TPA).

SECONDARY OUTCOMES:
Confirm the safety of intraventricular TPA. | 6 months
  Intrathecal TPA has been administered to many hundreds of patients world-wide, and continues to be widely used despite a paucity of strong evidence demonstrating efficacy. Thus, we believe the safety has been relatively well established. On the other hand, much of the existing data is observational and retrospective, and could therefore be vulnerable to reporting bias. Experience is more limited among patients who have been managed with endovascular coil embolization, such that our study will provide important additional safety information.
Assess feasibility of a future multi-center trial | 6 months
  By performing a single center, prospective, randomized, double-blind, placebo-controlled trial, we will be able to (1) Estimate the recruitment rate; (2) Establish whether clinicians can be successfully blinded to treatment allocation (TPA vs. placebo); (3) Ensure that clinicians will comply with a treatment protocol

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kramer, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada